CLINICAL TRIAL: NCT00139698
Title: A Phase III, Multicenter, Open-Label, Dose-Titrating, 16-Week Study Evaluating The Efficacy, Tolerability and Safety of Olmesartan Medoxomil 20 Mg and 40 Mg Alone or in Combination With 12.5 Mg to 25 Mg of Hydrochlorothiazide in Subjects With Mild to Moderate Essential Hypertension
Brief Title: Olmesartan Alone or in Combination With Hydrochlorothiazide in Subjects With Mild to Moderate Essential Hypertension
Acronym: OSCAR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A0021002
Record Dates: First submitted 2005-08-29; First posted 2005-08-31 (Estimated); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Essential Hypertension
MeSH Terms: conditions — Essential Hypertension | interventions — olmesartan; Hydrochlorothiazide

INTERVENTIONS:
Drug: olmesartan alone or in combination with hydrochlorothiazide

SUMMARY:
Efficacy, tolerability and safety of olmesartan alone or in combination with hydrochlorothiazide in the treatment of mild to moderate essential hypertension

ELIGIBILITY:
Inclusion Criteria:

* Subject has mild to moderate hypertension

Exclusion Criteria:

* History of secondary hypertension

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 410
Dates: Start 2005-09; Study Completion 2006-07

PRIMARY OUTCOMES:
Efficacy of olmesartan alone or in combination with hydrochlorothiazide in the treatment of mild to moderate essential hypertension

SECONDARY OUTCOMES:
Safety and tolerability of olmesartan alone or in combination with hydrochlorothiazide in the treatment of mild to moderate essential hypertension

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (27):
- Colombia (5):
  - Pfizer Investigational Site, Medellín, Antioquia
  - Pfizer Investigational Site, Barranquilla, Atlántico
  - Pfizer Investigational Site, Cartagena, Atlántico
  - Pfizer Investigational Site, Bogota, Cundinamarca
  - Pfizer Investigational Site, Cali, Valle del Cauca Department
- Ecuador (2):
  - Pfizer Investigational Site, Escobedo, Guayas
  - Pfizer Investigational Site, Quito, Pichincha
- Hong Kong (2):
  - Pfizer Investigational Site, NT
  - Pfizer Investigational Site, Shatin, NT
- Indonesia (2):
  - Pfizer Investigational Site, Jakarta
  - Pfizer Investigational Site, Surabaya
- Malaysia (2):
  - Pfizer Investigational Site, Seremban, Negeri Sembilan
  - Pfizer Investigational Site, Kuching, Sarawak
- Philippines (2):
  - Pfizer Investigational Site, San Juan City, National Capital Region
  - Pfizer Investigational Site, Quezon
- Pfizer Investigational Site, Singapore, Singapore
- Taiwan (3):
  - Pfizer Investigational Site, Guei-Shan Shiang, Tau-Yuan Shian
  - Pfizer Investigational Site, Kaohsiung City
  - Pfizer Investigational Site, Taipei
- Thailand (3):
  - Pfizer Investigational Site, Khet Rajathevee, Bangkok
  - Pfizer Investigational Site, Bangkok
  - Pfizer Investigational Site, Chiang Mai
- Turkey (Türkiye) (4):
  - Pfizer Investigational Site, Bornova/Izmir
  - Pfizer Investigational Site, Haseki/Istanbul
  - Pfizer Investigational Site, SÂ¿hhiye/Ankara
  - Pfizer Investigational Site, Sihhiye/Ankara
- Pfizer Investigational Site

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0021002&StudyName=Olmesartan+Alone+or+in+Combination+With+Hydrochlorothiazide+in+Subjects+With+Mild+to+Moderate+Essential+Hypertension